CLINICAL TRIAL: NCT05968755
Title: Leveraging Chatbot Technology to Improve PrEP Awareness and Uptake Among Black MSM in the Southern United States
Brief Title: Leveraging Chatbot to Improve PrEP in the Southern United States
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2000035242; 000 (Other: CTGTY)
Record Dates: First submitted 2023-05-22; First posted 2023-08-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: HIV Prevention; PrEP Awareness; PrEP Uptake

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: A chatbot designed to promote PrEP awareness and uptake for Black MSM
- Control group (Placebo Comparator)
  Interventions: Other: General educational messages

INTERVENTIONS:
Device: A chatbot designed to promote PrEP awareness and uptake for Black MSM — Participants in the intervention group will have access to a theory-informed (Self-Determination Theory) chatbot and receive an automated personalized question message (root-node message) from the chatbot. The root-node messages are questions written into the chatbot algorithms to initiate interactive communication with participants. In each round of the interactive communication, the chatbot will provide automated personalized PrEP-related information, autonomous motivation, and psychological needs based on Self-Determination Theory constructs.
  Arms: Intervention group
Other: General educational messages — Participants in the control group will received general education messages from a research assistant including healthy diet, exercise, and COVID-19 prevention. The frequency of contact will be pre-specified by participants in interviews prior to the RCT.
  Arms: Control group

SUMMARY:
The purpose of this study is to develop a chatbot intervention to promote PrEP awareness and uptake among Black men who have sex with men (MSM) in the Southern United States.

DETAILED DESCRIPTION:
In the United States (US), the epicenter of the HIV epidemic is in the South. The HIV-related death rate in the US South is high, but engagement with quality HIV prevention services and care is low. Although only 38% of the US population lives in the South, the region accounts for 51% of new HIV infections. Gay, bisexual, and other men who have sex with men (MSM) account for 60% of new infections among African Americans in the South. Black MSM are one of the most vulnerable groups to HIV transmission in the US. HIV testing and PrEP uptake in Black MSM, however, remain low (10%) due to multiple factors including stigma, sexual-orientation based discrimination and low PrEP awareness among Black MSM. Innovative strategies that motivate and provide guidance for PrEP among Black MSM in the US South are therefore urgently needed. Chatbot technology should be tested and implemented to help improve PrEP awareness and uptake in the US South. In this project, the investigators aim to develop and pilot test to assess the acceptability and feasibility of a chatbot for PrEP awareness and uptake relative to treatment as usual (control).

ELIGIBILITY:
Inclusion Criteria:

* Being cisgender Black male
* Being aged ≥ 18 years
* Having Internet access
* Speaking English
* Self-reporting condomless sex with another man in the past 6 months
* HIV negative or untested.

Exclusion Criteria:

* Having lived in the US South less than 3 months
* Having received antiretroviral therapy (ART) treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2026-03-28 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline PrEP awareness in 90 days | At baseline, 30 days, 60 days, and 90 days
  PrEP awareness will be measured as the proportion of participants who are aware of PrEP. Specifically, the investigators will collect PrEP awareness by asking participants standardized questions through a Qualtrics survey.
Change from baseline PrEP uptake in 90 days | At baseline, 30 days, 60 days, and 90 days
  PrEP uptake will be measured as the mean of the frequency of taking PrEP medication. Specifically, the investigators will collect PrEP uptake by asking participants through a Qualtrics survey if they have been taken PrEP at baseline and every 30 days. If participants respond that they have taken PrEP, the investigators will ask them the date and frequency of taking it and ask them to upload a photo of their PrEP for verification to reduce social desirability bias in responses.

SECONDARY OUTCOMES:
Change in Usability score | At baseline, 30 days, 60 days, and 90 days
  The usability score will be measured by the System Usability Scale, which is 5-point Likert scale consisted of 10 questions. Participants' scores range from 0 to 100. A score of 68 is average, below 68 is poor, above 68 is good, and above 80.3 is excellent.
Change in Recommendation score | At baseline, 30 days, 60 days, and 90 days
  The recommendation score will be calculated by a Net Promote Score, which measures MSM's likelihood to recommend the chatbot to other MSM friends. The score ranges from 0 to 10. The higher the score, the better the recommendation score.
Change in Acceptability score | At baseline, 30 days, 60 days, and 90 days
  Acceptability, defined as the extent to which the chatbot is suitable and satisfactory to MSM, will be measured using the standardized Customer Satisfaction Scale "How would you rate your overall satisfaction with the chatbot?" and a 5-point Likert question "How would you rate the likelihood of continuing to use the chatbot?"
Change in Practicality score | At baseline, 30 days, 60 days, and 90 days
  Practicality defined as the extent to which the chatbot provides real-time Self-Determination theory inputs, will be measured using a 5-point Likert question "How would you rate the overall quality of the chatbot?"
Change in Demand score | At baseline, 30 days, 60 days, and 90 days
  Demand, defined as the level of integration to which the chatbot fits into the MSM-preferred online platform, will be measured by the number of actual use documented on developer's platform.
Change in Adaptation score | At baseline, 30 days, 60 days, and 90 days
  Adaptation, defined as the extent to which the chatbot can be integrated into other social-networking apps, will be measured by asking "How likely would you use the chatbot if embedded on other apps?"

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Ni, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Care 4 U Community Health Center, Miami, Florida
  - Community Care Resources of FL (CCRSFL), Pembroke Pines, Florida
  - NAESM, Inc, Atlanta, Georgia
  - RAO Community Health, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. HIV and African American Gay and Bisexual Men. [cited 2022 August 4]; Available from: https://www.cdc.gov/hiv/group/msm/bmsm.html.
- [Background] Adeagbo O, Harrison S, Qiao S, Li X. Pre-Exposure Prophylaxis (PrEP) Uptake among Black Men Who Have Sex with Men (BMSM) in the Southern U.S. Int J Environ Res Public Health. 2021 Sep 15;18(18):9715. doi: 10.3390/ijerph18189715. PMID 34574652
- [Background] Watson RJ, Eaton LA, Maksut JL, Rucinski KB, Earnshaw VA. Links Between Sexual Orientation and Disclosure Among Black MSM: Sexual Orientation and Disclosure Matter for PrEP Awareness. AIDS Behav. 2020 Jan;24(1):39-44. doi: 10.1007/s10461-019-02696-1. PMID 31606770